CLINICAL TRIAL: NCT04037254
Title: Randomized Phase II Trial of Niraparib With Standard Combination Radiotherapy and Androgen Deprivation Therapy (ADT) in High Risk Prostate Cancer (With Initial Phase I) (NADIR*) *Randomized Phase II Trial of Niraparib With Standard Combination Androgen DeprIvation Therapy (ADT) and Radiotherapy in High Risk Prostate Cancer (With Initial Phase I)
Brief Title: Testing the Addition of a New Anti-Cancer Drug, Niraparib, to the Usual Treatment (Hormone and Radiation Therapy) for Prostate Cancer With a High Chance of Recurring
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: NRG Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NRG-GU007; NCI-2019-02260 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); NRG-GU007 (Other: NRG Oncology); NRG-GU007 (Other: CTEP); U10CA180868 (NIH)
Record Dates: First submitted 2019-07-26; First posted 2019-07-30 (Actual); Results first posted 2025-07-11 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: Prostate Adenocarcinoma; Stage IIC Prostate Cancer AJCC v8; Stage III Prostate Cancer AJCC v8; Stage IIIA Prostate Cancer AJCC v8; Stage IIIB Prostate Cancer AJCC v8; Stage IIIC Prostate Cancer AJCC v8; Stage IVA Prostate Cancer AJCC v8
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Gonadotropin-Releasing Hormone; Radiotherapy, Intensity-Modulated; niraparib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Phase I, Dose Level 1 (niraparib, GnRH, IMRT) (Experimental): Patients undergo standard of care GnRH agonist androgen suppression therapy for 24 months and concurrent niraparib PO QD* for the first 12 months. Beginning 8 weeks after starting niraparib, patients undergo standard of care IMRT 5 days per week for about 6-9 weeks depending on type of radiation therapy. Treatment is given in the absence of disease progression or unacceptable toxicity.
  *Niraparib dose level 1: 100 mg.
  Interventions: Biological: Gonadotrophin Releasing Hormone; Radiation: Intensity-Modulated Radiation Therapy; Drug: Niraparib
- Phase I, Dose Level 2 (niraparib, GnRH, IMRT) (Experimental): Patients undergo standard of care GnRH agonist androgen suppression therapy for 24 months and concurrent niraparib PO QD* for the first 12 months. Beginning 8 weeks after starting niraparib, patients undergo standard of care IMRT 5 days per week for about 6-9 weeks depending on type of radiation therapy. Treatment is given in the absence of disease progression or unacceptable toxicity.
  *Niraparib dose level 2: 100 mg during IMRT 200 mg otherwise.
  Interventions: Biological: Gonadotrophin Releasing Hormone; Radiation: Intensity-Modulated Radiation Therapy; Drug: Niraparib
- Phase I, Dose Level 3 (niraparib, GnRH, IMRT) (Experimental): Patients undergo standard of care GnRH agonist androgen suppression therapy for 24 months and concurrent niraparib PO QD* for the first 12 months. Beginning 8 weeks after starting niraparib, patients undergo standard of care IMRT 5 days per week for about 6-9 weeks depending on type of radiation therapy. Treatment given in the absence of disease progression or unacceptable toxicity.
  *Niraparib dose level 3: 200 mg.
  Interventions: Biological: Gonadotrophin Releasing Hormone; Radiation: Intensity-Modulated Radiation Therapy; Drug: Niraparib
- Phase II, Arm I (GnRH, IMRT) (Active Comparator): Patients undergo standard of care GnRH agonist androgen suppression therapy for 24 months. Beginning 8-28 weeks after starting GnRH agonist, patients undergo IMRT 5 days per week for about 6-9 weeks depending on type of radiation therapy. Treatment is given in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Gonadotrophin Releasing Hormone; Radiation: Intensity-Modulated Radiation Therapy
- Phase II, Arm II (niraparib, GnRH, IMRT) (Experimental): Patients undergo standard of care GnRH agonist androgen suppression therapy for 24 months and concurrent niraparib PO QD (phase I determined dose level) for the first 12 months. Beginning 8 weeks after starting niraparib, patients undergo standard of care IMRT 5 days per week for about 6-9 weeks depending on type of radiation therapy. Treatment is given in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Gonadotrophin Releasing Hormone; Radiation: Intensity-Modulated Radiation Therapy; Drug: Niraparib

INTERVENTIONS:
Biological: Gonadotrophin Releasing Hormone — Receive standard of care GnRH agonist androgen suppression therapy
  Other Names: AY-24031; D-His-6-Pro-8-NEt-LHRH; Follicle Stimulating Hormone-Releasing Factor; GN-RH; GnRH; Gonadoliberin; Gonadorelin; Gonadorelinum; gonadotropin-releasing hormone; Hoe- 471; LH-RF; LH-RH; LH/FSH-RF; LH/FSH-RH; LHRH; Luliberin; Luteinising Hormone-Releasing Factor; Luteinizing Hormone-Releasing Factor; Luteinizing Hormone-Releasing Hormone
Radiation: Intensity-Modulated Radiation Therapy — Undergo standard of care IMRT
  Other Names: IMRT; Intensity modulated radiation therapy (procedure); Intensity Modulated RT; Intensity-Modulated Radiotherapy; Radiation, Intensity-Modulated Radiotherapy
Drug: Niraparib — tablet
  Other Names: MK 4827; MK-4827; MK4827
  Arms: Phase I, Dose Level 1 (niraparib, GnRH, IMRT); Phase I, Dose Level 2 (niraparib, GnRH, IMRT); Phase I, Dose Level 3 (niraparib, GnRH, IMRT); Phase II, Arm II (niraparib, GnRH, IMRT)

SUMMARY:
This is a phase I-II trial to find the safety and activity of adding a new drug (neraparib) to the usual treatment (radiation combined with male hormone deprivation therapy) in lowering the chance of prostate cancer growing or returning. Niraparib is an inhibitor of PARP, an enzyme that helps repair deoxyribonucleic acid (DNA) when it becomes damaged. Blocking PARP may help keep cancer cells from repairing their damaged DNA, causing them to die. PARP inhibitors are a type of targeted therapy. Adding niraparib to the usual care may lower the chance of prostate cancer growing or returning.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To establish the preferred dose of niraparib in combination with radiation and antiandrogen therapy (ADT). (Phase I) II. To compare the disease-free state, defined as prostate specific antigen (PSA) remaining < 0.1 ng/ml at the end of ADT therapy in men with high risk prostate cancer treated with standard therapy with or without the addition of niraparib. (Phase IIR)

SECONDARY OBJECTIVES:

I. To further establish the safety and toxicity profile of standard treatment with radiation and androgen deprivation therapy specifically, two years from initiation of ADT, plus niraparib at the phase II dose.

II. To compare the overall survival, prostate cancer-specific survival, local/regional or distant progression, and distant metastatic disease rates of standard therapy with or without the addition of niraparib.

EXPLORATORY OBJECTIVE:

I. To identify genomic biomarkers of response to combination therapy with radiation, ADT and PARP inhibition.

OUTLINE: This is a phase I, dose-escalation study of niraparib, followed by a randomized phase II study.

PHASE I: Patients receive niraparib orally (PO) once daily (QD) and receive standard of care gonadotrophin releasing hormone (GnRH) agonist androgen suppression therapy. Treatment with niraparib continues for 12 months, and GnRH agonist therapy for 24 months in the absence of disease progression or unacceptable toxicity. Beginning 8 weeks after starting niraparib and GnRH agonist, patients undergo standard of care intensity-modulated radiation therapy (IMRT) 5 days per week for about 6-9 weeks, depending on type of radiation therapy given, in the absence of disease progression or unacceptable toxicity. Patients also undergo magnetic resonance imaging (MRI) on study.

PHASE II: Patients are randomized to 1 of 2 arms:

ARM I: Patients undergo standard of care GnRH agonist androgen suppression therapy for 24 months in the absence of disease progression or unacceptable toxicity. Beginning 8-28 weeks after starting GnRH agonist, patients undergo IMRT 5 days per week for about 6-9 weeks depending on type of radiation therapy given in the absence of disease progression or unacceptable toxicity. Patients also undergo MRI on study.

ARM II: Patients undergo standard of care GnRH agonist androgen suppression therapy for 24 months, and niraparib PO QD for 12 months in the absence of disease progression or unacceptable toxicity. Beginning 8 weeks after starting niraparib, patients undergo standard of care IMRT 5 days per week for about 6-9 weeks depending on type of radiation therapy given in the absence of disease progression or unacceptable toxicity. Patients also undergo MRI on study.

After completion of study treatment, patients are followed up every 6 months for 3 years, then annually for 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed (within 180 days prior to registration) adenocarcinoma of the prostate at high risk for recurrence as determined by the following criteria, according to American Joint Committee on Cancer (AJCC) 8th edition:

  * Phase I enrollment

    * Gleason >= 9, PSA =< 150 ng/mL, any T-stage
  * Phase II enrollment

    * Gleason >= 9, PSA =< 150 ng/mL, any T-stage
    * Gleason 8, PSA < 20 ng/mL, and >= T2
    * Gleason 8, PSA >= 20-150 ng/mL, any T-stage
    * Gleason 7, PSA >= 20-150 ng/mL, any T-stage
* No distant metastases as evaluated by:

  * Bone scan 90 days prior to registration
  * Lymph node assessment by computed tomography (CT) or magnetic resonance (MR) of pelvis or nodal sampling within 90 days prior to registration (Please note: Lymph nodes will be considered negative [N0] if they are < 1.5 cm short axis)
* History/physical examination within 90 days prior to registration
* Age >= 18
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1 within 180 days prior to registration
* Pretreatment serum PSA, obtained prior to any androgen suppression therapy and within 180 days of registration
* Phase I patients: Prior androgen suppression for prostate cancer is not allowed prior to registration
* Phase II patients: Prior androgen suppression for prostate cancer is allowed =< 45 days prior to registration
* Hemoglobin >= 9.0 g/dL (within 90 days prior to registration)
* Platelets >= 100,000 cells/mm^3 (within 90 days prior to registration)
* Absolute neutrophil count (ANC) >= 1.5 x 10^9/L (within 90 days prior to registration)
* Serum creatinine =<1.5 x upper limit of normal (ULN) OR a calculated creatinine clearance >= 30 mL/min estimated using Cockcroft-Gault equation (within 90 days prior to registration)
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) =< 3.0 x ULN (within 90 days prior to registration)
* Serum albumin >= 3 g/dL (within 90 days prior to registration)
* Serum potassium >= 3.5 mmol/L (within 90 days prior to registration)
* Serum total bilirubin =< 1.5 x ULN or direct bilirubin =< 1 x ULN (Note: in subjects with Gilberts syndrome, if total bilirubin is > 1.5 x ULN, measure direct and indirect bilirubin, and if direct bilirubin is =< 1.5 x ULN, subject may be eligible) (within 90 days prior to registration)
* Men of child-producing potential must be willing to consent to use effective contraception while on treatment and for at least 3 months afterwards
* The patient or a legally authorized representative must provide study-specific informed consent prior to study entry

Exclusion Criteria:

* PSA > 150 ng/mL
* Definitive clinical or radiologic evidence of metastatic disease
* Pathologically positive lymph nodes or nodes > 1.5 cm short axis on CT or MR imaging
* Prior radical prostatectomy, cryosurgery for prostate cancer, or bilateral orchiectomy for any reason
* Any active malignancy within 2 years of study registration that may alter the course of prostate cancer treatment
* Prior systemic therapy for prostate cancer; note that prior therapy for a different cancer is allowable
* Prior radiotherapy, including brachytherapy, to the region of the prostate that would result in overlap of radiation therapy fields
* Current treatment with first generation anti-androgens (bicalutamide, nilutamide, flutamide). For patients enrolled to phase II, if prior anti-androgens were administered, a washout period of >= 30 days is required prior to enrollment
* Severe, active co-morbidity, defined as follows:

  * Unstable angina and/or congestive heart failure requiring hospitalization within the last 6 months
  * Transmural myocardial infarction within the last 6 months
  * Acute bacterial or fungal infection requiring intravenous antibiotics at the time of registration
  * Uncontrolled acquired immune deficiency syndrome (AIDS) based upon current Centers for Disease Control and Prevention (CDC) definition
  * Presence of uncontrolled hypertension (persistent systolic blood pressure [BP] >=160 mmHg or diastolic BP >= 100 mmHg). Subjects with a history of hypertension are allowed, provided that BP is controlled to within these limits by anti-hypertensive treatment
* Prior allergic reaction to the drugs involved in this protocol (including known allergies, hypersensitivity or intolerance to the excipients of niraparib)
* Human immunodeficiency virus (HIV) positive with CD4 count < 200 cells/microliter

  * Note that patients who are HIV positive are eligible, provided they have a CD4 count >= 200 cells/microliter within 90 days prior to registration. Patients receiving treatment with highly active antiretroviral therapy (HAART) will not be eligible due to concern for radiosensitization
  * Note also that HIV testing is not required for eligibility for this protocol. This exclusion criterion is necessary because the treatments involved in this protocol may be affected by these drugs
* Any history or current diagnosis of myelodysplastic syndrome (MDS)/acute myeloid leukemia (AML)
* Prior or current treatment with PARP inhibitor

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2019-10-08 (Actual); Primary Completion 2024-07-01 (Actual); Study Completion 2025-09-26 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: M. D Michaelson, Principal Investigator — NRG Oncology
Locations (95):
- United States (94):
  - Banner MD Anderson Cancer Center, Gilbert, Arizona
  - University of Arizona Cancer Center-Orange Grove Campus, Tucson, Arizona
  - University of Arizona Cancer Center-North Campus, Tucson, Arizona
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Cedars Sinai Medical Center, Los Angeles, California
  - Fremont - Rideout Cancer Center, Marysville, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - City of Hope Upland, Upland, California
  - Helen F Graham Cancer Center, Newark, Delaware
  - Medical Oncology Hematology Consultants PA, Newark, Delaware
  - George Washington University Medical Center, Washington D.C., District of Columbia
  - Grady Health System, Atlanta, Georgia
  - Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia
  - Emory Saint Joseph's Hospital, Atlanta, Georgia
  - CTCA at Southeastern Regional Medical Center, Newnan, Georgia
  - Alton Memorial Hospital, Alton, Illinois
  - Northwestern University, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - University of Kansas Cancer Center, Kansas City, Kansas
  - University of Kansas Cancer Center-Overland Park, Overland Park, Kansas
  - University of Kansas Hospital-Westwood Cancer Center, Westwood, Kansas
  - University of Maryland/Greenebaum Cancer Center, Baltimore, Maryland
  - Central Maryland Radiation Oncology in Howard County, Columbia, Maryland
  - UM Baltimore Washington Medical Center/Tate Cancer Center, Glen Burnie, Maryland
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - McLaren Cancer Institute-Bay City, Bay City, Michigan
  - Henry Ford Cancer Institute-Downriver, Brownstown, Michigan
  - McLaren Cancer Institute-Clarkston, Clarkston, Michigan
  - Henry Ford Macomb Hospital-Clinton Township, Clinton Township, Michigan
  - Henry Ford Medical Center-Fairlane, Dearborn, Michigan
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Weisberg Cancer Treatment Center, Farmington Hills, Michigan
  - McLaren Cancer Institute-Flint, Flint, Michigan
  - Singh and Arora Hematology Oncology PC, Flint, Michigan
  - Karmanos Cancer Institute at McLaren Greater Lansing, Lansing, Michigan
  - Mid-Michigan Physicians-Lansing, Lansing, Michigan
  - McLaren Cancer Institute-Lapeer Region, Lapeer, Michigan
  - McLaren Cancer Institute-Macomb, Mount Clemens, Michigan
  - Henry Ford Medical Center-Columbus, Novi, Michigan
  - McLaren Cancer Institute-Northern Michigan, Petoskey, Michigan
  - McLaren-Port Huron, Port Huron, Michigan
  - Henry Ford Macomb Health Center - Shelby Township, Shelby, Michigan
  - Henry Ford West Bloomfield Hospital, West Bloomfield, Michigan
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Siteman Cancer Center at Saint Peters Hospital, City of Saint Peters, Missouri
  - Siteman Cancer Center at West County Hospital, Creve Coeur, Missouri
  - University of Kansas Cancer Center - North, Kansas City, Missouri
  - University of Kansas Cancer Center - Lee's Summit, Lee's Summit, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Siteman Cancer Center-South County, St Louis, Missouri
  - Benefis Sletten Cancer Institute, Great Falls, Montana
  - AtlantiCare Health Park-Cape May Court House, Cape May Court House, New Jersey
  - AtlantiCare Surgery Center, Egg Harbor, New Jersey
  - Rutgers New Jersey Medical School, Newark, New Jersey
  - Holy Name Hospital, Teaneck, New Jersey
  - Roswell Park Cancer Institute, Buffalo, New York
  - The New York Hospital Medical Center of Queens, Flushing, New York
  - Highland Hospital, Rochester, New York
  - University of Rochester, Rochester, New York
  - Stony Brook University Medical Center, Stony Brook, New York
  - Summa Health System - Akron Campus, Akron, Ohio
  - Summa Health System - Barberton Campus, Barberton, Ohio
  - University of Cincinnati Cancer Center-UC Medical Center, Cincinnati, Ohio
  - Case Western Reserve University, Cleveland, Ohio
  - Summa Health Medina Medical Center, Medina, Ohio
  - University of Cincinnati Cancer Center-West Chester, West Chester, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Christiana Care Health System-Concord Health Center, Chadds Ford, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Penn State Milton S Hershey Medical Center, Hershey, Pennsylvania
  - Geisinger Medical Oncology-Lewisburg, Lewisburg, Pennsylvania
  - Lewistown Hospital, Lewistown, Pennsylvania
  - Eastern Regional Medical Center, Philadelphia, Pennsylvania
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania
  - UPMC-Shadyside Hospital, Pittsburgh, Pennsylvania
  - Geisinger Wyoming Valley/Henry Cancer Center, Wilkes-Barre, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Prisma Health Cancer Institute - Faris, Greenville, South Carolina
  - Saint Francis Cancer Center, Greenville, South Carolina
  - Prisma Health Cancer Institute - Eastside, Greenville, South Carolina
  - Self Regional Healthcare, Greenwood, South Carolina
  - Prisma Health Cancer Institute - Greer, Greer, South Carolina
  - Prisma Health Cancer Institute - Seneca, Seneca, South Carolina
  - West Virginia University Healthcare, Morgantown, West Virginia
  - Froedtert Menomonee Falls Hospital, Menomonee Falls, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
  - Zablocki Veterans Administration Medical Center, Milwaukee, Wisconsin
  - Drexel Town Square Health Center, Oak Creek, Wisconsin
  - ProHealth Oconomowoc Memorial Hospital, Oconomowoc, Wisconsin
  - UW Cancer Center at ProHealth Care, Waukesha, Wisconsin
  - Froedtert West Bend Hospital/Kraemer Cancer Center, West Bend, Wisconsin
- Arthur J E Child Comprehensive Cancer Centre, Calgary, Alberta, Canada

RESULTS

PARTICIPANT FLOW:
Groups:
- Phase I, Dose Level 1 (DL1) (Niraparib, GnRH, IMRT): Patients undergo standard of care gonadotrophin releasing hormone (GnRH) agonist androgen suppression therapy for 24 months, and niraparib PO QD* for 12 months in the absence of disease progression or unacceptable toxicity. Beginning 8 weeks after starting niraparib, patients undergo standard of care intensity-modulated radiation therapy (IMRT) 5 days per week for about 6-9 weeks depending on type of radiation therapy given in the absence of disease progression or unacceptable toxicity.
  *niraparib dose level 1: 100 mg.
- Phase I, Dose Level 2 (DL2) (Niraparib, GnRH, IMRT): Patients undergo standard of care GnRH agonist androgen suppression therapy for 24 months, and niraparib PO QD* for 12 months in the absence of disease progression or unacceptable toxicity. Beginning 8 weeks after starting niraparib, patients undergo standard of care IMRT 5 days per week for about 6-9 weeks depending on type of radiation therapy given in the absence of disease progression or unacceptable toxicity.
  *niraparib dose level 2: 100 mg during IMRT 200 mg all other time.
- Phase I, Dose Level 3 (DL3) (Niraparib, GnRH, IMRT): Patients undergo standard of care GnRH agonist androgen suppression therapy for 24 months, and niraparib PO QD* for 12 months in the absence of disease progression or unacceptable toxicity. Beginning 8 weeks after starting niraparib, patients undergo standard of care IMRT 5 days per week for about 6-9 weeks depending on type of radiation therapy given in the absence of disease progression or unacceptable toxicity.
  *niraparib dose level 3: 200 mg.
- Phase II, Arm I (GnRH, IMRT): Patients undergo standard of care GnRH agonist androgen suppression therapy for 24 months in the absence of disease progression or unacceptable toxicity. Beginning 8-28 weeks after starting GnRH agonist, patients undergo IMRT 5 days per week for about 6-9 weeks depending on type of radiation therapy given in the absence of disease progression or unacceptable toxicity. Patients also undergo MRI on study.
- Phase II, Arm II (Niraparib, GnRH, IMRT): Patients undergo standard of care GnRH agonist androgen suppression therapy for 24 months, and niraparib PO QD (phase I determined dose level) for 12 months in the absence of disease progression or unacceptable toxicity. Beginning 8 weeks after starting niraparib, patients undergo standard of care IMRT 5 days per week for about 6-9 weeks depending on type of radiation therapy given in the absence of disease progression or unacceptable toxicity.
Period: Overall Study
Arm/Group | Phase I, Dose Level 1 (DL1) (Niraparib, GnRH, IMRT) | Phase I, Dose Level 2 (DL2) (Niraparib, GnRH, IMRT) | Phase I, Dose Level 3 (DL3) (Niraparib, GnRH, IMRT) | Phase II, Arm I (GnRH, IMRT) | Phase II, Arm II (Niraparib, GnRH, IMRT)
Started | 7 | 7 | 8 | 0 | 0
Eligible and Evaluable | 6 | 5 | 6 | 0 | 0
Completed | 6 | 5 | 6 | 0 | 0
Not Completed | 1 | 2 | 2 | 0 | 0
Not completed — Protocol Violation | 1 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0 | 0
Not completed — Delayed or incomplete treatment | 0 | 2 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Eligible and evaluable phase I participants. (Phase II component will not open.)
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase I, Dose Level 1 (Niraparib, GnRH, IMRT) | Phase I, Dose Level 2 (Niraparib, GnRH, IMRT) | Phase I, Dose Level 3 (Niraparib, GnRH, IMRT) | Total
Number analyzed (Participants) | 6 | 5 | 6 | 17
Age, Continuous [Median (Full Range); unit: years] | 72.5 [61 to 78] | 74 [64 to 78] | 71 [60 to 79] | 72 [60 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 6 | 5 | 6 | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 6 | 5 | 6 | 17
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 1 | 2
  White | 5 | 5 | 5 | 15
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
T-Stage [Count of Participants; unit: Participants] — Tumor stage per the American Joint Committee on Cancer (AJCC) X8h ed. refers to the size and/or extent of the main tumor. The higher the number after the T, the larger the tumor or the more it has grown into nearby tissues.
  * T1: The tumor is too small to be felt or seen on imaging;
  * T2: The tumor is confined within the prostate;
  * T3: The tumor has grown outside the prostate;
  * T4: The tumor has spread to nearby tissues other than the seminal vesicles.
  Participants
    T1 | 0 | 1 | 1 | 2
    T2 | 6 | 2 | 3 | 11
    T3 | 0 | 1 | 2 | 3
    T4 | 0 | 1 | 0 | 1
N-Stage [Count of Participants; unit: Participants] — Regional lymph nodes staging per American Joint Committee on Cancer (AJCC) 8th ed. refers to the number and/or extent of spread of lymph nodes that contain cancer:
  * N0: The cancer has not spread to any nearby lymph nodes;
  * N1: The cancer has spread to one or more nearby lymph nodes
  Participants
    N0 | 6 | 5 | 6 | 17
    N1 | 0 | 0 | 0 | 0
Gleason score [Count of Participants; unit: Participants] — Gleason score describes prostate cancer based on how abnormal the cancer cells in a biopsy sample look under a microscope. Cells are scored 1-5 with 1 indicating "low-grade" looking similar to normal cells and 5 indicating "high-grade" barely resembling normal cells due to mutation. A pathologist assigns a Gleason grade to the first and second most predominant patterns in the biopsy. The two grades are added together to calculate the Gleason score (between 2 and 10). Cancers with lower scores tend to be less aggressive, while cancers with higher scores end to be more aggressive.
  Participants
    9 | 5 | 5 | 6 | 16
    10 | 1 | 0 | 0 | 1
Baseline Prostate-specific antigen (PSA) [Count of Participants; unit: Participants] — Prostate-specific antigen (PSA) is a protein made by the prostate gland and found in the blood. PSA blood levels may be higher than normal in men who have prostate cancer, benign prostatic hyperplasia (BPH), or infection or inflammation of the prostate gland, and are often used to monitor patients who have been treated for prostate cancer to see if their cancer has recurred.
  Participants
    PSA < 20 ng/mL | 5 | 5 | 6 | 16
    PSA ≥ 20-150 ng/mL | 1 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Disease-free Until Completion of Treatment (2 Years From Start of ADT)
Description: Participants will be considered disease-free if their PSA values remain below 0.1 ng/ml until the completion of treatment. The proportion of patients disease-free at 24 months were to be compared in the two treatment arms using a non-continuity-corrected chi-square test. PSA levels will be assessed prior to the start of RT, at the end of RT, and every three months for 24 months. all PSA values obtained up to and including the two-year landmark must be < 0.1 ng/ml. Patients who die prior to two years from prostate cancer will be counted as failures. Patients who die from causes other than prostate cancer will be considered non-evaluable for the primary endpoint. Patients still under follow-up but who have a missing PSA value at two years or more than two missing values prior to two years will also be counted as failures.
Time Frame: Baseline to completion of treatment (two years from start of ADT)
Population: Eligible and evaluable phase II participants followed for two years after start of ADT. The study did/will not advance to the phase II component.
Arm/Group | Phase II, Arm I (GnRH, IMRT) | Phase II, Arm II (Niraparib, GnRH, IMRT)
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Percent of Participants Alive (Overall Survival)
Description: Survival rates were to be estimated using the Kaplan-Meier method and the treatment arms were to be compared using a log-rank test.
Time Frame: From baseline to death or last follow-up, analyzed after phase II participants have been followed for two years, which was expected to occur 3.5 years from start of phase II component.
Population: Eligible phase II participants. The study did/will not advance to the phase II component.
Arm/Group | Phase II, Arm I (GnRH, IMRT) | Phase II, Arm II (Niraparib, GnRH, IMRT)
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Percentage of Participants With Prostate Cancer Deaths (Prostate Cancer-specific Survival)
Description: Prostate cancer death rates were to be estimated using the cumulative incidence method, treating deaths due to other causes as competing risks. The treatment arms were to be compared using the Fine-Gray test
Time Frame: From baseline to death or last follow-up, analyzed after all phase II participants have been followed for two years, which was expected to occur 3.5 years from start of phase II component.
Population: Eligible phase II participants. The study did/will not advance to the phase II component.
Arm/Group | Phase II, Arm I (GnRH, IMRT) | Phase II, Arm II (Niraparib, GnRH, IMRT)
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Percentage of Participants With Pathologic Complete Response (pCR) at Two Years
Description: Complete response was to be determined by a12-core biopsy. Treatment arms were to be compared using a chi-square test.
Time Frame: At two years
Population: Eligible phase II participants with 12-core biopsy at 24 months. The study did/will not advance to the phase II component.
Arm/Group | Phase II, Arm I (GnRH, IMRT) | Phase II, Arm II (Niraparib, GnRH, IMRT)
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Percentage of Participants With Local/Regional or Distant Progression
Description: Progression rates were to be estimated using the cumulative incidence method, treating deaths as competing risks. The treatment arms were to be compared using the Fine-Gray test
Time Frame: From baseline to local/regional or distant progression, death, or last follow-up, whichever occurs first, analyzed after all phase II participants have been followed for two years, which was expected to occur 3.5 years from start of phase II component.
Population: Eligible phase II participants. The study did/will not advance to the phase II component.
Arm/Group | Phase II, Arm I (GnRH, IMRT) | Phase II, Arm II (Niraparib, GnRH, IMRT)
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Percentage of Participants With Distant Metastases
Description: Distant metastases rates were to be estimated using the cumulative incidence method, treating death as a competing risk. The treatment arms were to be compared using the Fine-Gray test
Time Frame: From baseline to distant metastasis, death, or last follow-up, analyzed after all phase II participants have been followed for two years, which was expected to occur 3.5 years from start of phase II component.
Population: Eligible phase II participants. The study did not and will not advance to the phase II component.
Arm/Group | Phase II, Arm I (GnRH, IMRT) | Phase II, Arm II (Niraparib, GnRH, IMRT)
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Percentage of Participants Alive Without Biochemical Progression (Biochemical Progression-free Survival)
Description: Biochemical progression is defined as PSA ≥ 2 ng/ml over the nadir PSA, the presence of local, regional, or distant recurrence, or death from prostate cancer. Biochemical progression-free survival rates were to be estimated using the Kaplan-Meier method and the treatment arms were to be compared using a log-rank test.
Time Frame: From baseline to biochemical progression or last follow-up, analyzed after all phase II participants have been followed for two years, which was expected to occur 3.5 years from start of phase II component.
Population: Eligible phase II participants. The study did/will not advance to the phase II component.
Arm/Group | Phase II, Arm I (GnRH, IMRT) | Phase II, Arm II (Niraparib, GnRH, IMRT)
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Number of Participants by Highest Grade Adverse Event Reported
Description: Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 grades adverse event severity as follows: 1 = mild, 2 = moderate, 3 = severe, 4 = life-threatening, 5 = death related to adverse event. Summary data is provided in this outcome measure; see Adverse Events Module for specific adverse event data. Adverse events were to be categorized as early (within 90 days of completion of radiotherapy) or late (more than 90 days after the completion of radiotherapy).The number of participants per grade was to be compared between the arms for early, late, and all adverse events using chi-square or Fisher exact tests
Time Frame: From baseline to last follow-up, analyzed after all phase II participants have been followed for two years, which was expected to occur 3.5 years from start of phase II component.
Population: Eligible phase II participants. The study did not and will not advance to the phase II component.
Arm/Group | Phase II, Arm I (GnRH, IMRT) | Phase II, Arm II (Niraparib, GnRH, IMRT)
Number analyzed (Participants) | 0 | 0

9. Other Pre Specified Outcome: Maximum Tolerated Dose (MTD) of Niraparib/ Preferred Niraparib Dose for Phase II Component
Description: MTD was determined using the classic 3+3 design to determine the safety of each dose level (DL) from the number of participants with dose limiting toxicities (DLTs), starting with DL1. The highest DL deemed safe was to be considered the MTD. The timing of the 3-patient cohorts took into account the previously established safety of concurrent ADT and 200 mg niraparib and the need to more clearly establish the safety of niraparib concurrent with RT. A DLT is defined as any treatment-related gastrointestinal or genitourinary grade 3 or higher AE lasting > 1 week, despite maximal medical interventions, and any treatment-related grade 4 AEs lasting > 1 week. Relationship to treatment was determined by the responsible clinician. Study chairs reviewed possible DLTs for final determination.
  Niraparib dose level (mg PO QD) definitions [First 8 weeks with ADT, 6-8 weeks with ADT and RT, remaining time of the 12 months]:
  * DL1: 100, 100, 100
  * DL2: 200, 100, 200
  * DL3: 200, 200, 200
Time Frame: From start of combined ADT and niraparib to six months
Population: Eligible and evaluable phase I participants.
Measure: Number; unit: Dose level
Groups:
- All Participants: Patients undergo standard of care GnRH agonist androgen suppression therapy for 24 months, and niraparib PO QD* for 12 months in the absence of disease progression or unacceptable toxicity. Beginning 8 weeks after starting niraparib, patients undergo standard of care IMRT 5 days per week for about 6-9 weeks depending on type of radiation therapy given in the absence of disease progression or unacceptable toxicity.
  Niraparib dose level 1: 100 mg. Niraparib dose level 2: 100 mg during IMRT, 200 mg all other time. Niraparib dose level 3: 200 mg.
Arm/Group | All Participants
Number analyzed (Participants) | 17
Dose level | 3

10. Other Pre Specified Outcome: Number of Participants Who Experienced Dose-limiting Toxicities (DLT)
Description: A DLT is defined as any treatment-related gastrointestinal or genitourinary grade 3 or higher AE lasting > 1 week, despite maximal medical interventions, and any treatment-related grade 4 AEs lasting > 1 week. Relationship to treatment was determined by the responsible clinician. Study chairs reviewed possible DLTs for final determination.
Time Frame: From start of combined ADT and niraparib to six months
Population: Eligible and evaluable phase I participants.
Measure: Count of Participants; unit: Participants
Groups:
- Phase I, Dose Level 1 (Niraparib, GnRH, IMRT): Patients undergo standard of care GnRH agonist androgen suppression therapy for 24 months, and niraparib PO QD* for 12 months in the absence of disease progression or unacceptable toxicity. Beginning 8 weeks after starting niraparib, patients undergo standard of care IMRT 5 days per week for about 6-9 weeks depending on type of radiation therapy given in the absence of disease progression or unacceptable toxicity.
  *niraparib dose level 1: 100 mg.
- Phase I, Dose Level 2 (Niraparib, GnRH, IMRT): Patients undergo standard of care GnRH agonist androgen suppression therapy for 24 months, and niraparib PO QD* for 12 months in the absence of disease progression or unacceptable toxicity. Beginning 8 weeks after starting niraparib, patients undergo standard of care IMRT 5 days per week for about 6-9 weeks depending on type of radiation therapy given in the absence of disease progression or unacceptable toxicity.
  *niraparib dose level 2: 100 mg during IMRT 200 mg all other time.
- Phase I, Dose Level 3 (Niraparib, GnRH, IMRT): Patients undergo standard of care GnRH agonist androgen suppression therapy for 24 months, and niraparib PO QD* for 12 months in the absence of disease progression or unacceptable toxicity. Beginning 8 weeks after starting niraparib, patients undergo standard of care IMRT 5 days per week for about 6-9 weeks depending on type of radiation therapy given in the absence of disease progression or unacceptable toxicity.
  *niraparib dose level 3: 200 mg.
Arm/Group | Phase I, Dose Level 1 (Niraparib, GnRH, IMRT) | Phase I, Dose Level 2 (Niraparib, GnRH, IMRT) | Phase I, Dose Level 3 (Niraparib, GnRH, IMRT)
Number analyzed (Participants) | 6 | 5 | 6
Participants | 0 | 0 | 0

11. Other Pre Specified Outcome: Percentage of Participants With Gene Alterations Detected by Targeted Exome Sequencing
Description: The percentage of patients with baseline or post-therapy alterations in targeted genes would be reported and the association between the occurrence of alterations and clinical outcomes would be assessed.
Time Frame: From baseline to death or last follow-up, analyzed after all participants have been followed for two years and gene mutation data produced
Population: Eligible phase II participants with gene alteration data. The study did not and will not advance to the phase II component.
Arm/Group | Phase II, Arm I (GnRH, IMRT) | Phase II, Arm II (Niraparib, GnRH, IMRT)
Number analyzed (Participants) | 0 | 0

12. Other Pre Specified Outcome: Percentage of Participants With Gene Expression Determined by High-density Affymetrix Oligonucleotide Array to Profile the Transcriptome of Tumor Samples
Description: The percentage of participants with baseline or post-therapy gene expression and the association between the occurrence of alterations and clinical outcomes would be assessed.
Time Frame: From baseline to death or last follow-up, analyzed after all participants have been followed for two years and gene expression data generated.
Population: Eligible phase II participants with gene expression data. The study did not and will not advance to the phase II component.
Arm/Group | Phase II, Arm I (GnRH, IMRT) | Phase II, Arm II (Niraparib, GnRH, IMRT)
Number analyzed (Participants) | 0 | 0

13. Other Pre Specified Outcome: Percentage of Participants With Single Nucleotide Polymorphisms From Whole Blood Samples
Description: The percentage of patients with baseline or post-therapy polymorphism would be reported and the association between the occurrence of alterations and clinical outcomes would be assessed.
Time Frame: From baseline to death or last follow-up, analyzed after all participants have been followed for two years and polymorphism data generated.
Population: Eligible phase II participants with polymorphism data. The study did not and will not advance to the phase II component.
Arm/Group | Phase II, Arm I (GnRH, IMRT) | Phase II, Arm II (Niraparib, GnRH, IMRT)
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: From baseline to last follow-up. Maximum follow-up was 4.6 years.
Description: All-cause mortality and adverse events were assessed in eligible and evaluable phase I participants. The study did not and will not advance to the phase II component.
Arm/Group | Phase I, Dose Level 1 (Niraparib, GnRH, IMRT) | Phase I, Dose Level 2 (Niraparib, GnRH, IMRT) | Phase I, Dose Level 3 (Niraparib, GnRH, IMRT)
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/5 | 0/6
Serious Adverse Events (participants affected / at risk) | 3/6 | 3/5 | 3/6
Other Adverse Events (participants affected / at risk) | 6/6 | 5/5 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase I, Dose Level 1 (Niraparib, GnRH, IMRT) (N=6) | Phase I, Dose Level 2 (Niraparib, GnRH, IMRT) (N=5) | Phase I, Dose Level 3 (Niraparib, GnRH, IMRT) (N=6)
ANEMIA (Blood and lymphatic system disorders) | 0 | 1 | 0
ATRIAL FIBRILLATION (Cardiac disorders) | 1 | 0 | 0
CHEST PAIN - CARDIAC (Cardiac disorders) | 1 | 0 | 0
PALPITATIONS (Cardiac disorders) | 1 | 0 | 0
LIMBAL STEM CELL DEFICIENCY (Eye disorders) | 1 | 0 | 0
CONSTIPATION (Gastrointestinal disorders) | 1 | 0 | 0
DIARRHEA (Gastrointestinal disorders) | 2 | 0 | 0
HEMORRHOIDAL HEMORRHAGE (Gastrointestinal disorders) | 1 | 0 | 0
NAUSEA (Gastrointestinal disorders) | 1 | 0 | 0
PROCTITIS (Gastrointestinal disorders) | 1 | 1 | 0
RECTAL HEMORRHAGE (Gastrointestinal disorders) | 1 | 0 | 0
RECTAL PAIN (Gastrointestinal disorders) | 1 | 0 | 0
SMALL INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 0 | 1 | 0
PAIN (General disorders) | 1 | 0 | 0
ABDOMINAL INFECTION (Infections and infestations) | 0 | 1 | 0
COVID (Infections and infestations) | 1 | 0 | 0
URINARY TRACT INFECTION (Infections and infestations) | 0 | 0 | 1
LYMPHOCYTE COUNT DECREASED (Investigations) | 0 | 0 | 1
NEUTROPHIL COUNT DECREASED (Investigations) | 0 | 0 | 1
WHITE BLOOD CELL DECREASED (Investigations) | 0 | 0 | 1
HYPERGLYCEMIA (Metabolism and nutrition disorders) | 1 | 0 | 1
HYPOKALEMIA (Metabolism and nutrition disorders) | 0 | 0 | 1
SEIZURE (Nervous system disorders) | 0 | 1 | 0
DYSURIA (Renal and urinary disorders) | 1 | 0 | 0
NOCTURIA (Renal and urinary disorders) | 0 | 0 | 1
URINARY URGENCY (Renal and urinary disorders) | 1 | 0 | 0
SINUS CONGESTION (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
YEAST INFECTION (R) GROIN (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
HOT FLASHES (Vascular disorders) | 1 | 0 | 0
THROMBOEMBOLIC EVENT (Vascular disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase I, Dose Level 1 (Niraparib, GnRH, IMRT) (N=6) | Phase I, Dose Level 2 (Niraparib, GnRH, IMRT) (N=5) | Phase I, Dose Level 3 (Niraparib, GnRH, IMRT) (N=6)
ANEMIA (Blood and lymphatic system disorders) | 5 | 2 | 5
DECREASED HEMATOCRIT (Blood and lymphatic system disorders) | 1 | 0 | 0
DECREASED MEAN CORPUSCULAR HEMOGLOBIN CONCENTRATION (Blood and lymphatic system disorders) | 1 | 0 | 0
DECREASED TOTAL PROTEIN (Blood and lymphatic system disorders) | 1 | 0 | 0
ELEVATED BLOOD UREA NITROGEN (Blood and lymphatic system disorders) | 1 | 0 | 0
EOSINOPHILIA (Blood and lymphatic system disorders) | 0 | 1 | 0
RED BLOOD CELL DECREASED (Blood and lymphatic system disorders) | 1 | 0 | 0
ATRIAL FIBRILLATION (Cardiac disorders) | 0 | 1 | 0
CHEST PAIN - CARDIAC (Cardiac disorders) | 2 | 0 | 0
SINUS TACHYCARDIA (Cardiac disorders) | 1 | 0 | 0
EAR PAIN (Ear and labyrinth disorders) | 1 | 0 | 0
VERTIGO (Ear and labyrinth disorders) | 1 | 0 | 0
HYPERTHYROIDISM (Endocrine disorders) | 0 | 0 | 1
ABDOMINAL PAIN (Gastrointestinal disorders) | 0 | 0 | 1
BLOATING (Gastrointestinal disorders) | 1 | 0 | 0
CONSTIPATION (Gastrointestinal disorders) | 3 | 3 | 2
DIARRHEA (Gastrointestinal disorders) | 4 | 1 | 3
DRY MOUTH (Gastrointestinal disorders) | 1 | 1 | 1
DYSPEPSIA (Gastrointestinal disorders) | 0 | 1 | 1
FLATULENCE (Gastrointestinal disorders) | 1 | 0 | 0
GLUTEN AND LACTOSE INTOLERANCE (Gastrointestinal disorders) | 1 | 0 | 0
HEMORRHOIDAL HEMORRHAGE (Gastrointestinal disorders) | 1 | 0 | 1
HEMORRHOIDS (Gastrointestinal disorders) | 1 | 0 | 0
NAUSEA (Gastrointestinal disorders) | 0 | 1 | 3
PROCTITIS (Gastrointestinal disorders) | 0 | 1 | 0
RECTAL HEMORRHAGE (Gastrointestinal disorders) | 0 | 0 | 1
RECTAL MUCOSITIS (Gastrointestinal disorders) | 0 | 1 | 0
TENESMUS (Gastrointestinal disorders) | 0 | 0 | 1
VOMITING (Gastrointestinal disorders) | 0 | 0 | 1
CHILLS (General disorders) | 0 | 1 | 0
EDEMA LIMBS (General disorders) | 1 | 0 | 0
FATIGUE (General disorders) | 3 | 5 | 5
FLU LIKE SYMPTOMS (General disorders) | 0 | 1 | 0
GENERALIZED EDEMA (General disorders) | 0 | 0 | 1
INJECTION SITE REACTION (General disorders) | 1 | 0 | 1
PAIN (General disorders) | 1 | 0 | 0
SINUS INFECTION (Infections and infestations) | 0 | 0 | 1
SINUSITIS (Infections and infestations) | 1 | 0 | 0
SKIN INFECTION (Infections and infestations) | 0 | 0 | 1
UPPER RESPIRATORY INFECTION (Infections and infestations) | 1 | 0 | 0
URINARY TRACT INFECTION (Infections and infestations) | 0 | 0 | 1
FALL (Injury, poisoning and procedural complications) | 3 | 0 | 0
SPINAL FRACTURE (Injury, poisoning and procedural complications) | 0 | 0 | 1
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 1 | 0 | 1
ALKALINE PHOSPHATASE INCREASED (Investigations) | 0 | 0 | 1
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 2 | 1 | 1
BLOOD BILIRUBIN INCREASED (Investigations) | 1 | 0 | 1
BLOOD LACTATE DEHYDROGENASE INCREASED (Investigations) | 0 | 0 | 1
CREATININE INCREASED (Investigations) | 1 | 0 | 1
LYMPHOCYTE COUNT DECREASED (Investigations) | 3 | 1 | 5
NEUTROPHIL COUNT DECREASED (Investigations) | 1 | 0 | 1
PLATELET COUNT DECREASED (Investigations) | 2 | 0 | 1
WEIGHT GAIN (Investigations) | 2 | 0 | 1
WEIGHT LOSS (Investigations) | 1 | 1 | 1
WHITE BLOOD CELL DECREASED (Investigations) | 1 | 0 | 3
ANOREXIA (Metabolism and nutrition disorders) | 1 | 1 | 1
HYPERCALCEMIA (Metabolism and nutrition disorders) | 0 | 1 | 0
HYPERGLYCEMIA (Metabolism and nutrition disorders) | 1 | 0 | 1
HYPERKALEMIA (Metabolism and nutrition disorders) | 1 | 1 | 1
HYPERTRIGLYCERIDEMIA (Metabolism and nutrition disorders) | 1 | 0 | 1
HYPOALBUMINEMIA (Metabolism and nutrition disorders) | 1 | 0 | 0
HYPOCALCEMIA (Metabolism and nutrition disorders) | 1 | 0 | 0
HYPOKALEMIA (Metabolism and nutrition disorders) | 1 | 0 | 0
HYPONATREMIA (Metabolism and nutrition disorders) | 1 | 0 | 1
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 1 | 0 | 2
ARTHRITIS (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
BACK PAIN (Musculoskeletal and connective tissue disorders) | 2 | 1 | 2
GENERALIZED MUSCLE WEAKNESS (Musculoskeletal and connective tissue disorders) | 2 | 0 | 1
MUSCLE CRAMP (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
ATAXIA (Nervous system disorders) | 1 | 0 | 0
COGNITIVE DISTURBANCE (Nervous system disorders) | 0 | 1 | 0
DIZZINESS (Nervous system disorders) | 2 | 2 | 0
DYSESTHESIA (Nervous system disorders) | 1 | 0 | 0
DYSGEUSIA (Nervous system disorders) | 0 | 1 | 0
HEADACHE (Nervous system disorders) | 1 | 0 | 2
PERIPHERAL SENSORY NEUROPATHY (Nervous system disorders) | 1 | 0 | 1
TREMOR (Nervous system disorders) | 1 | 0 | 0
DEPRESSION (Psychiatric disorders) | 2 | 0 | 0
INSOMNIA (Psychiatric disorders) | 0 | 3 | 1
DYSURIA (Renal and urinary disorders) | 2 | 0 | 3
HEMATURIA (Renal and urinary disorders) | 0 | 2 | 2
NOCTURIA (Renal and urinary disorders) | 1 | 3 | 1
PROTEINURIA (Renal and urinary disorders) | 1 | 0 | 0
RADIATION CYSTITIS (Renal and urinary disorders) | 0 | 0 | 1
STOP AND START URINATION (Renal and urinary disorders) | 0 | 1 | 0
STRAIN TO BEGIN URINATION (Renal and urinary disorders) | 0 | 1 | 0
URINARY FREQUENCY (Renal and urinary disorders) | 5 | 4 | 3
URINARY HESITANCY (Renal and urinary disorders) | 0 | 0 | 2
URINARY INCONTINENCE (Renal and urinary disorders) | 3 | 0 | 0
URINARY RETENTION (Renal and urinary disorders) | 1 | 2 | 1
URINARY TRACT OBSTRUCTION (Renal and urinary disorders) | 1 | 1 | 0
URINARY URGENCY (Renal and urinary disorders) | 3 | 2 | 3
WEAK STREAM (Renal and urinary disorders) | 0 | 1 | 1
ERECTILE DYSFUNCTION (Reproductive system and breast disorders) | 1 | 1 | 0
COUGH (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1
DYSPNEA (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 0
NASAL CONGESTION (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
SINUS CONGESTION (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
DRY SKIN (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
HYPERHIDROSIS (Skin and subcutaneous tissue disorders) | 1 | 1 | 1
PRURITUS (Skin and subcutaneous tissue disorders) | 0 | 0 | 2
RASH ACNEIFORM (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
RASH MACULO-PAPULAR (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
VERY SMALL AMOUNT OF BLOOD ON TISSUE WHEN WIPES AT TIMES (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
HOT FLASHES (Vascular disorders) | 4 | 4 | 5
HYPERTENSION (Vascular disorders) | 1 | 0 | 1
PERIPHERAL ISCHEMIA (Vascular disorders) | 0 | 1 | 0

LIMITATIONS AND CAVEATS:
This study closed accrual permanently without proceeding to the phase II component because the standard of care for prostate cancer in this population substantially evolved and incorporation of the new standard would have required a much larger sample size. Therefore, only phase I results can be reported, appearing as "other pre-specified" outcome measures because although listed as a primary objective in the protocol, they are not explicitly listed as primary or secondary statistical endpoints.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI's are required to abide by the sponsor's publication guidelines which require review by coauthors and subsequent review and approval by the sponsor.

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-05-24): https://cdn.clinicaltrials.gov/large-docs/54/NCT04037254/Prot_SAP_000.pdf
  • Informed Consent Form (2022-05-24): https://cdn.clinicaltrials.gov/large-docs/54/NCT04037254/ICF_001.pdf